CLINICAL TRIAL: NCT06753968
Title: The Role of Natural Orifice Specimen Extraction Surgery (NOSES) in Treating Right-sided Colon Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, China (Other)
Responsible Party: Principal Investigator, Haitao Zhou, Professor Haitao Zhou, National Cancer Center, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOSES for right hemicolectomy
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Colon Cancer
Keywords: colon cancer; totallly laparoscopic right hemicolectomy; natural orifice specimen extraction surgery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Right Hemicolectomy With Transrectal/transvaginal Specimen Extraction (NOSES) (Experimental): The NOSES group employs two distinct methods for specimen extraction, both of which have been thoroughly outlined in previous studies. The first method, transvaginal extraction, begins with the irrigation and disinfection of the vagina, followed by a transverse incision in the posterior fornix. The assistant then utilizes oval forceps to carefully extract the specimen bag through the incision, which is subsequently closed with continuous full-thickness sutures, using barbed sutures to ensure secure closure. The second method, transrectal extraction, similarly begins with irrigation of the rectum using a dilute iodine solution, followed by a longitudinal incision along the anterior wall of the upper rectum. The specimen, along with the protective sleeve, is then removed using oval forceps, and the incision is closed with a continuous full-layer running suture once the specimen has been completely extracted.
  Interventions: Procedure: Laparoscopic Right Hemicolectomy With Transrectal/transvaginal Specimen Extraction (NOSES)
- Totally Laparoscopic Right Hemicolectomy (TLRH) (Active Comparator): Totally Laparoscopic Right Hemicolectomy (TLRH), which involves performing intracorporeal anastomosis and specimen extraction through a small abdominal incision, enhances the benefits of minimally invasive surgery In the TLRH group, following the stapled side-to-side anastomosis, a small horizontal incision is made about 2 to 3 cm above the symphysis pubis, at the junction of the pubic hairline, to allow for specimen removal.
  Interventions: Procedure: Totally laparoscopic right hemicolectomy (TLRH)

INTERVENTIONS:
Procedure: Laparoscopic Right Hemicolectomy With Transrectal/transvaginal Specimen Extraction (NOSES) — Transvaginal extraction, begins with the irrigation and disinfection of the vagina, followed by a transverse incision in the posterior fornix. The assistant then utilizes oval forceps to carefully extract the specimen bag through the incision, which is subsequently closed with continuous full-thickness sutures, using barbed sutures to ensure secure closure. Similarly, transrectal extraction begins with irrigation of the rectum using a dilute iodine solution, followed by a longitudinal incision along the anterior wall of the upper rectum. The specimen, along with the protective sleeve, is then removed using oval forceps, and the incision is closed with a continuous full-layer running suture once the specimen has been completely extracted.
  Arms: Laparoscopic Right Hemicolectomy With Transrectal/transvaginal Specimen Extraction (NOSES)
Procedure: Totally laparoscopic right hemicolectomy (TLRH) — Totally laparoscopic right hemicolectomy (TLRH), which involves performing intracorporeal anastomosis and specimen extraction through a small abdominal incision, further enhances the benefits of minimally invasive surgery. In the TLRH group, following the stapled side-to-side anastomosis, a small horizontal incision is made about 2 to 3 cm above the symphysis pubis, at the junction of the pubic hairline, to allow for specimen removal.
  Arms: Totally Laparoscopic Right Hemicolectomy (TLRH)

SUMMARY:
The purpose of this study is to investigate the short-term and long-term outcomes between natural orifice specimen extraction surgery (NOSES) and totally laparoscopic right hemicolectomy (TLRH). The hypothesis is that NOSES could achieve good short-term and oncological outcomes for right colon cancer patients.

DETAILED DESCRIPTION:
This study is a retrospective clinical study. We reviewed collected data from all patients who underwent laparoscopic curative resection for stage I-III right-sided colon cancer between January 2018 and January 2023. A total of consecutive 115 patients who underwent laparoscopic resection with transvaginal or transrectal specimen extraction were identified as the NOSES group. To establish a comparative cohort, 234 patients who underwent totally laparoscopic right hemicolectomy (TLRH) during the same period were selected. The purpose of this study is to investigate the short-term and long-term outcomes between NOSES and TLRH. The hypothesis is that NOSES could promote postoperative recovery, reduce incision-related complications with comaprable long-term oncological outcomes when compared with TLRH.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven colon carcinoma;
2. Imaging diagnosis of T1-3 colon cancer;
3. The tumor located in the cecum, ascending colon, or colonic hepatic flexure;
4. Written informed consent;

Exclusion Criteria:

1. Complete intestinal obstruction;
2. Hepatitis activity and peripheral neuropathy (such as peripheral neuritis, pseudo meningitis, motor neuritis, and sensory impairment);
3. Significant organ dysfunction or other significant diseases, including clinically relevant coronary artery disease, cardiovascular disease, or myocardial infarction within the 12 months before enrollment; severe neurological or psychiatric history; severe infection; active disseminated intravascular coagulation;
4. Pregnancy or breastfeeding;
5. Alcohol abuse or drug addiction;
6. Concurrent uncontrolled medical condition;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
The rate of postoperative complications | up to 30 days
  The rate of postoperative complications = patients with any postoperative complications/all cases.

SECONDARY OUTCOMES:
Operating time | up to 1 days
  Operating time = The Operative time was defined as the time first skin incision was made to final skin closure
The time of first flatus | up to 5 days
  The time of first flatus = The time of first flatus reported by patients
Postoperative hospitalization | up to 30 days
  Postoperative hospitalization = the number of nights from surgery to discharge

OTHER OUTCOMES:
Estimated blood loss | up to 1 days
  Estimated blood loss = The sum of the blood in the suction canister (the total volume after subtracting the amount of irrigation fluid used) and the segment of increased weight of swabs used during operation phase (1 ml of blood is about weighs 1g)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Beijing, Beijing 100000, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Participants' data are only allowed to be used for the analysis of this study and are not authorized to be shared with other researchers.

REFERENCES:
- [Result] Li XW, Wang CY, Zhang JJ, Ge Z, Lin XH, Hu JH. Short-term efficacy of transvaginal specimen extraction for right colon cancer based on propensity score matching: A retrospective cohort study. Int J Surg. 2019 Dec;72:102-108. doi: 10.1016/j.ijsu.2019.07.025. Epub 2019 Jul 27. PMID 31362128